CLINICAL TRIAL: NCT00862940
Title: A 1-year Randomised, Double-blind Placebo-controlled Study to Evaluate the Effects of Memantine on Rate of Brain Atrophy in Patients With Alzheimer's Disease
Brief Title: A Clinical Study Evaluating the Effects of Memantine on Brain Atrophy in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10112; 2004-002614-10 (EudraCT Number)
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Alzheimer's Disease
Keywords: Memantine; Neuroimaging; MRI; Brain atrophy
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Experimental)
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — 10 mg tablets twice daily
  Other Names: Ebixa®
  Arms: Memantine
Drug: Placebo — Tablets twice daily
  Arms: Placebo

SUMMARY:
Pre-clinical studies have demonstrated that memantine can decrease the neuronal toxicity associated with excessive glutamate release and calcium overload in neurons. Previous studies have shown that memantine helps to treat the symptoms of Alzheimer's Disease (AD). In AD, the rate of brain tissue loss, or atrophy, is faster than in normal aging and this seems to go hand in hand with some of the symptoms of the disease. This suggests that memantine treatment in AD could provide both symptomatic improvement and neuro-protective effects. The purpose of this study was to show whether memantine, in addition to providing symptomatic benefits, can slow the rate of brain atrophy as assessed using magnetic resonance imaging (MRI) technology.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the effects of memantine on the rate of brain atrophy compared to placebo in patients with AD (moderate severity) over a 1-year period. This was a multinational, randomised, double-blind, parallel-group, placebo-controlled, fixed-dose study (20 mg memantine). The study also included secondary imaging, cognitive and behavioural measures.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients at least 50 years of age with a current diagnosis of probable AD of moderate severity (MMSE score between 12 and 20, inclusive) consistent with NINCDS-ADRDA criteria and MRI scans
* Patients must have had a knowledgeable and reliable caregiver to accompany them to all clinic visits during the study
* Patients were either on or off existing acetylcholinesterase inhibitor (AChEI) treatment provided that the treatment had been initiated >6 months prior to screening, had stabilised with respect to dose for >3 months, and remained fixed during the entire study. AChEI treatment could not be initiated or modified during the study

Exclusion Criteria:

* The patient had evidence of clinically significant active disease (including recent myocardial infarction and uncompensated congestive heart failure [NYHA II-IV])
* The patient had evidence of any clinically significant neurodegenerative disease or neurological disorder other than AD
* The patient was contraindicated for MRI

Other protocol-defined inclusion and exclusion criteria applied.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2005-09; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Result] Wilkinson D, Fox NC, Barkhof F, Phul R, Lemming O, Scheltens P. Memantine and brain atrophy in Alzheimer's disease: a 1-year randomized controlled trial. J Alzheimers Dis. 2012;29(2):459-69. doi: 10.3233/JAD-2011-111616. PMID 22269160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from each investigator's outpatient clinic.
Pre-assignment Details: After a 3-week run-in period during which MRI scans were performed, the patients were randomised to either placebo or memantine and stratified according to AChEI treatment. Memantine-treated patients started with 5 mg/day and were uptitrated by 5 mg/day every week for 4 weeks. The target dose of 20 mg/day was administered from the start of Week 4.
Period: Overall Study
Arm/Group | Memantine 10 mg Tablets Twice Daily | Placebo Tablets Twice Daily
Started | 133 | 144
Completed | 103 | 114
Not Completed | 30 | 30
Not completed — Adverse Event | 15 | 12
Not completed — Lack of Efficacy | 1 | 3
Not completed — Protocol Violation | 2 | 5
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Non-compliance | 4 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative or other reason(s) | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine 10 mg Tablets Twice Daily | Placebo Tablets Twice Daily | Total
Number analyzed (Participants) | 133 | 144 | 277
Age Continuous [Mean (Standard Deviation); unit: years] | 73.7 (8.8) | 74.4 (7.7) | 74.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 75 | 158
  Male | 50 | 69 | 119
Controlled Oral Word Association Test (COWAT): Baseline Efficacy Scores [Mean (Standard Deviation); unit: Number of words] — COWAT: Verbal fluency test. The patient was asked to, during 1 minute, generate as many words as possible beginning with three pre-specified letters. The total score was calculated as the sum of acceptable words generated, with higher scores indicating lower cognitive impairment.
  Number of words | 19.7 (10.3) | 19.2 (8.8) | 19.4 (9.6)
Category Fluency Test (CFT): Baseline Efficacy Scores [Mean (Standard Deviation); unit: Number of words] — CFT: The patient was asked to, during 1 minute, say aloud as many different words as possible from the categories animals and fruits. The total score was calculated as the number of appropriate words generated, with higher scores indicating lower cognitive impairment.
  Number of words | 13.5 (5.8) | 13.3 (5.9) | 13.4 (5.9)
ADAS-cog-Orientation Test (ADAS-cog-OT): Baseline Efficacy Scores [Mean (Standard Deviation); unit: Points] — ADAS-cog-OT: A subscale of the ADAS-cog test with 8 questions and designed to determine how well oriented the patient is with regard to time and place. The total score was calculated as 8 minus the total number of correct answers, with higher scores indicating greater cognitive impairment.
  Points | 4.2 (1.6) | 4.0 (1.7) | 4.1 (1.7)
Stroop Interference Test - Incongruent (SIT-I): Baseline Efficacy Scores [Mean (Standard Deviation); unit: Seconds] — SIT-I: A test to demonstrate the reaction time. Names of colours are printed in a different ink than the colour named. The time taken to complete the test was recorded, as was the number of errors. The more time spent and the higher number of errors indicates lower reaction time.
  Seconds | 170.3 (60.4) | 176.4 (56.7) | 173.4 (58.5)
Stroop Interference Test - Congruent (SIT-C): Baseline Efficacy Scores [Mean (Standard Deviation); unit: Seconds] — SIT-C: A test to demonstrate the reaction time. Names of colours are printed in the same ink as the colours named. The time taken to complete the test was recorded, as was the number of errors. The more time spent and the higher number of errors indicates lower reaction time.
  Seconds | 70.5 (49.1) | 68.8 (41.7) | 69.6 (45.4)
Mini Mental State Examination (MMSE): Baseline Efficacy Scores [Mean (Standard Deviation); unit: Points] — MMSE: Brief, structured examination of mental status that assesses orientation, memory, attention, naming, comprehension, and praxis. The range is 0 to 30, with a lower score indicating a worse mental state.
  Points | 16.9 (2.4) | 17.0 (2.4) | 16.9 (2.4)
Neuropsychiatric Inventory (NPI): Baseline Efficacy Scores [Mean (Standard Deviation); unit: Points] — NPI: A scale specifically developed to assess behavioural disturbances in patients with dementia. It is based on responses from the caregiver. The range is 0 to 120, with higher score reflecting higher frequency and severity of the disturbances.
  Points | 13.1 (12.8) | 12.8 (12.4) | 13.0 (12.6)
Magnetic Resonance Imaging (MRI) Descriptives [Mean (Standard Deviation); unit: mL; mm^3]
  Total Brain Volume (TBV) | 957.9 (103.3) | 968.9 (108.3) | 963.6 (105.8)
  Hippocampal Volume (HCV) | 5063.0 (1014.3) | 5107.6 (836.7) | 5086.1 (924.9)

OUTCOME MEASURES:

1. Primary Outcome: Total Brain Atrophy Rate Estimated Using Brain Boundary Shift Integral (BBSI)
Description: Measures direct changes in total brain volume per visit interval (screening to Week 4, 42, or 52 or from Week 4 to Week 42 or 52)
Time Frame: Baseline to 1 year
Population: FAS-MRI: Full-analysis set for all patients in the all-patients-treated set (APTS) who had at least one valid MRI scan >=6 months after initiation of investigational medicinal product (IMP). The FAS (full analysis set, efficacy set) replaces the intention-to-treat (ITT) concept used in older terminology.
Measure: Mean (Standard Error); unit: mL/year
Arm/Group | Memantine 10 mg Tablets Twice Daily | Placebo Tablets Twice Daily
Number analyzed (Participants) | 110 | 118
mL/year | 15.24 (0.97) | 15.32 (0.91)
Statistical Analysis 1: Comparison: Memantine 10 mg Tablets Twice Daily vs Placebo Tablets Twice Daily; Linear mixed model relating direct change in brain volume (BBSI) to time and its interaction with treatment group. This model additionally includes a time-by-AChEI group interaction as a fixed effect; Test type: Superiority or Other; p = 0.9754, Mixed Models Analysis; Adjusted mean difference = -0.04, 95% CI 2-sided [-2.60 to 2.52], Standard Error of Mean 1.30

2. Secondary Outcome: Changes in Total Hippocampal Volume (HCV)
Description: Estimated mean changes in total HCV
Time Frame: Baseline to 1 year
Population: FAS-MRI
Measure: Mean (Standard Deviation); unit: mm^3/year
Arm/Group | Memantine 10 mg Tablets Twice Daily | Placebo Tablets Twice Daily
Number analyzed (Participants) | 95 | 109
mm^3/year | -218 (182) | -220 (171)
Statistical Analysis 1: Comparison: Memantine 10 mg Tablets Twice Daily vs Placebo Tablets Twice Daily; Mixed model repeated measurements (MMRM) with unstructured covariance including time, time-by-treatment, visit, pre-treatment HCV, and AChEI group; Test type: Superiority or Other; p = 0.842, MMRM; Adjusted mean difference = -3.50, 95% CI 2-sided [-38.04 to 31.04], Standard Error of Mean 17.52

3. Secondary Outcome: Cognitive and Behavioural Outcomes: Controlled Oral Word Association Test (COWAT) Total Score
Description: Adjusted mean change from baseline on cognitive and behavioural scores. COWAT: Verbal fluency test. The patient was asked to, during 1 minute, generate as many words as possible beginning with three pre-specified letters. The total score was calculated as the sum of acceptable words generated, with higher scores indicating lower cognitive impairment
Time Frame: Baseline to 1 year
Population: FAS, observed cases (OC)
Measure: Least Squares Mean (Standard Error); unit: Scale scores
Arm/Group | Memantine 10 mg Tablets Twice Daily | Placebo Tablets Twice Daily
Number analyzed (Participants) | 106 | 114
Scale scores | 0.78 (0.71) | -0.90 (0.69)
Statistical Analysis 1: Comparison: Memantine 10 mg Tablets Twice Daily vs Placebo Tablets Twice Daily; Test type: Superiority or Other; p = 0.034, MMRM — The p-value represents the difference from placebo for COWAT at Week 52 (MMRM); Mean Difference (Final Values) = 1.68, 95% CI 2-sided [0.13 to 3.23], Standard Error of Mean 0.79

4. Secondary Outcome: Cognitive and Behavioural Outcomes: Mini Mental State Examination (MMSE) Total Score
Description: Adjusted mean change from baseline on cognitive and behavioural scores. MMSE: Brief, structured examination of mental status that assesses orientation, memory, attention, naming, comprehension, and praxis. The range is 0 to 30, with a lower score indicating a worse mental state
Time Frame: Baseline to 1 year
Population: FAS, OC
Measure: Least Squares Mean (Standard Error); unit: Scale scores
Arm/Group | Memantine 10 mg Tablets Twice Daily | Placebo Tablets Twice Daily
Number analyzed (Participants) | 108 | 114
Scale scores | -0.50 (0.45) | -0.74 (0.44)
Statistical Analysis 1: Comparison: Memantine 10 mg Tablets Twice Daily vs Placebo Tablets Twice Daily; Test type: Superiority or Other; p = 0.602, MMRM — The p-value represents the difference from placebo for MMSE at Week 52 (MMRM); Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.67 to 1.15], Standard Error of Mean 0.46

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Memantine 10 mg Tablets Twice Daily | Placebo Tablets Twice Daily
Serious Adverse Events (participants affected / at risk) | 17/133 | 20/144
Other Adverse Events (participants affected / at risk) | 46/133 | 36/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine 10 mg Tablets Twice Daily (N=133) | Placebo Tablets Twice Daily (N=144)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (5) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia [gs] (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 8 (9)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pacemaker generated rhythm (Surgical and medical procedures) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer [gs] (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Social stay hospitalisation (Social circumstances) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine 10 mg Tablets Twice Daily (N=133) | Placebo Tablets Twice Daily (N=144)
Agitation (Psychiatric disorders) | 7 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 10 (11)
Dizziness (Nervous system disorders) | 11 (11) | 4 (8)
Fall (Injury, poisoning and procedural complications) | 8 (9) | 9 (10)
Headache (Nervous system disorders) | 9 (11) | 7 (8)
Urinary tract infection (Infections and infestations) | 7 (8) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and H. Lundbeck A/S. Manuscripts and abstracts must be sent to H. Lundbeck A/S at least one month prior to submission for publication or presentation.